CLINICAL TRIAL: NCT02682927
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled Trial of Two Fixed Doses of ZX008 (Fenfluramine Hydrochloride) Oral Solution as an Adjunctive Therapy in Children and Young Adults With Dravet Syndrome
Brief Title: A Trial of Two Fixed Doses of ZX008 (Fenfluramine HCl) in Children and Young Adults With Dravet Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zogenix International Limited, Inc., a subsidiary of Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZX008-1501; ZX008-1502 (Other: Zogenix International Limited, Inc., a subsidiary of Zogenix, Inc.); NCT02826863 (obsolete NCT alias)
Record Dates: First submitted 2016-02-05; First posted 2016-02-17 (Estimated); Results first posted 2022-10-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Dravet Syndrome; Seizure Disorder
Keywords: seizure; tonic-atonic; clonic; epilepsy; myoclonic; encephalopathy
MeSH Terms: conditions — Epilepsies, Myoclonic; Epilepsy; Seizures; Brain Diseases | interventions — Fenfluramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ZX008 - 0.8 mg/kg/day (Experimental): ZX008 (fenfluramine HCl) is supplied as an oral solution in concentrations of 1.25, 2.5, and 5 mg/mL. ZX008 will be administered twice a day (BID) in equally divided doses with food.
  Interventions: Drug: ZX008 (Fenfluramine Hydrochloride)
- ZX008 - 0.2 mg/kg/day (Experimental): ZX008 (fenfluramine HCl) is supplied as an oral solution in concentrations of 1.25, 2.5, and 5 mg/mL. ZX008 will be administered twice a day (BID) in equally divided doses with food.
  Interventions: Drug: ZX008 (Fenfluramine Hydrochloride)
- Matching Placebo (Placebo Comparator): Placebo will be administered twice a day (BID) in equally divided doses with food.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: ZX008 (Fenfluramine Hydrochloride) — ZX008 drug product is an oral aqueous solution of fenfluramine hydrochloride buffered to pH 5. The product is sugar free and is intended to be compatible with a ketogenic diet.
  Arms: ZX008 - 0.2 mg/kg/day; ZX008 - 0.8 mg/kg/day
Drug: Matching Placebo — Placebo solution for ZX008. The product is sugar free and is intended to be compatible with a ketogenic diet.
  Arms: Matching Placebo

SUMMARY:
Study 1 and Study 3 are the prospective, merged analyses of 2 identical double-blind, placebo-controlled studies, ZX008-1501 and ZX008-1502, to assess the efficacy, safety, and pharmacokinetics of ZX008 when used as adjunctive therapy in pediatric and young adult subjects with Dravet syndrome. Study 1501 and Study 1502 were conducted in parallel; Study 1501 was conducted at approximately 30 study sites in North America; Study 1502 was conducted at approximately 30 study sites in Europe, Asia and Australia. Upon completion of the Baseline Period after initial Screening and Baseline charting of seizure frequency, subjects who qualified for the studies were randomized (1:1:1) in a double-blind manner to receive either 1 of 2 doses of ZX008 (0.2 mg/kg/day or 0.8 mg/kg/day; maximum dose: 30 mg/day) or placebo. Randomization was stratified by age group (< 6 years, ≥6 to 18 years) to achieve balance across treatment arms, with the target of 25% of subjects in each age group. All subjects were titrated to their randomized dose over a 14-day Titration Period. Following titration, subjects continued treatment at their randomly assigned dose over a 12-week Maintenance Period. Subjects exiting the study underwent a 2-week taper, unless they enrolled in a follow-on study. Subjects were followed for post-study safety monitoring.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or non-pregnant, non-lactating female, age 2 to 18 years, inclusive as of the day of the Screening Visit.
* Clinical diagnosis of Dravet syndrome, where convulsive seizures are not completely controlled by current antiepileptic drugs.
* Must have a minimum # of convulsive seizures per 4-week period for past 12 weeks prior to screening.
* All medications or interventions for epilepsy must be stable for at least 4 weeks prior to screening and expected to remain stable throughout the study.
* No cardiovascular or cardiopulmonary abnormality based on ECHO, ECG or physical examination.
* Parent/caregiver is willing and able to be compliant with diary completion, visit schedule and study drug accountability.

Key Exclusion Criteria:

* Pulmonary arterial hypertension.
* Current or past history of cardiovascular or cerebrovascular disease, such as cardiac valvulopathy, myocardial infarction or stroke.
* Current or past history of glaucoma.
* Moderate or severe hepatic impairment.
* Receiving concomitant therapy with: anorectic agents; monoamine-oxidase inhibitors; medications that act via serotonin including serotonin reuptake inhibitors; atomoxetine, or other centrally-acting noradrenergic agonist; or cyproheptadine.
* Currently receiving or has received stiripentol in the past 21 days prior to Screening.
* Currently taking carbamazepine, oxcarbamazepine, eslicarbazepine, phenobarbital, or phenytoin, or has taken any of these within the past 30 days.
* Positive result on tetrahydrocannabinol (THC) or cannabidiol (CBD) test at the Screening Visit.
* A clinically significant medical condition,that would interfere with study participation, collection of study data, or pose a risk to the subject.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 262 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (55):
- United States (19):
  - Phoenix Children's, Phoenix, Arizona
  - Center for Neurosciences - Tucson, Tucson, Arizona
  - Rady Children's Hospital San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - The Children's Hospital Colorado, Aurora, Colorado
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Miami Children's Hospital Brain Institute, Miami, Florida
  - Neurology and Epilepsy Research Center, Orlando, Florida
  - Panda Neurology, Atlanta, Georgia
  - Children's Hospital of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
- Australia (3):
  - Melbourne Brain Centre Austin Hospital, Melbourne
  - Children's Health Queensland Hospital and Health Service at Lady Cilento Children's Hospital, South Brisbane
  - The Children's Hospital Westmead Dept. of Neurology and Neurosurgery, Westmead
- Universitair Ziekenhuis Antwerpen, Antwerp, Belgium
- Canada (2):
  - British Columbia Children's Hospital BCCH, Vancouver, British Columbia
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal
- Danish National Epilepsy Centre, Dianalund, Denmark
- French Ref centre Necker Hospital Paris, Paris, France
- Germany (8):
  - Epilepsiezentrum / Neuropädiatrie Hedwig-von-Rittberg-Zentrum Für Kinder und Jugendliche, Berlin
  - Krankenhaus Mara Epilepsie-Zentrum Bethel, Bielefeld
  - Epilepsiezentrum Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Jena Klinik fuer Kinder- und Jugendmedizin Neuropaediatrie, Jena
  - Klinik für Neuropädiatrie Universitätsklinikum Schleswig Holstein Campus Kiel, Kiel
  - Kleinwachau Saechsisches Epilepsiezentrum Radeberggemeinnuetzige GmbH, Radeberg
  - Universitaetsklinik fuer Kinder- und Jugendmedizin Abteilung III, Tübingen
  - Schoen Klinik Vogtareuth Neuropaediatrie und Neurologische Rehabilitation, Epilepsiezentrum fuer Kinder und Jugendlische,Tagesklinik fuer Neuropaediatrie, Vogtareuth
- Italy (7):
  - AOU Anna Meyer, Florence
  - Istituto Pediatrico Giannina Gaslini Dipartimento di Neurologia, Genova
  - A.O Carlo Poma, Mantova
  - Instituto Neurologica Carlo Besta, Milan
  - Ospedale Fatebenefratelli e Oftalmico, Milan
  - U.O. Neurologia Dipartimento di Neuroscienze Ospedale Pediatrico Bambino Gesù, IRCS, Roma
  - Ospedal Policlinico Giambattista Rossi diBorga Roma, Verona
- Japan (4):
  - Okayama University Hospital, Okayama, Okayama-ken
  - Saitama Children's Medical Center, Saitama-shi, Saitama
  - National Epilepsy Center Shizuoka Institute, Shizuoka, Shizuoka
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
- Spain (3):
  - Hospital Sant Joande Déu, Barcelona
  - Hospital Ruber Internacional Primera Planta Servicio de Neurologia, Madrid
  - Clinica Universitaria de Navarra Fase 4. Segunda planta, Consulta de Pediatria, Pamplona
- United Kingdom (6):
  - Birmingham Children Hospital, Birmingham
  - Institute of Neurosciences Queens Elizabeth University Hospital, Glasgow
  - Alder Hey Hospital, Liverpool
  - Evelina Hospital, London
  - Great Ormonnd Street Hospital for Children NHS Foundation Trust, London
  - Sheffield Children's Hospital, Sheffield

REFERENCES:
- [Result] Sullivan J, Lagae L, Cross JH, Devinsky O, Guerrini R, Knupp KG, Laux L, Nikanorova M, Polster T, Talwar D, Ceulemans B, Nabbout R, Farfel GM, Galer BS, Gammaitoni AR, Lock M, Agarwal A, Scheffer IE; FAiRE DS Study Group. Fenfluramine in the treatment of Dravet syndrome: Results of a third randomized, placebo-controlled clinical trial. Epilepsia. 2023 Oct;64(10):2653-2666. doi: 10.1111/epi.17737. Epub 2023 Aug 17. PMID 37543865
- [Derived] Cross JH, Galer BS, Gil-Nagel A, Devinsky O, Ceulemans B, Lagae L, Schoonjans AS, Donner E, Wirrell E, Kothare S, Agarwal A, Lock M, Gammaitoni AR. Impact of fenfluramine on the expected SUDEP mortality rates in patients with Dravet syndrome. Seizure. 2021 Dec;93:154-159. doi: 10.1016/j.seizure.2021.10.024. Epub 2021 Nov 2. PMID 34768178
- [Derived] Sullivan J, Specchio N, Devinsky O, Auvin S, Perry MS, Strzelczyk A, Gil-Nagel A, Dai D, Galer BS, Gammaitoni AR. Fenfluramine significantly reduces day-to-day seizure burden by increasing number of seizure-free days and time between seizures in patients with Dravet syndrome: A time-to-event analysis. Epilepsia. 2022 Jan;63(1):130-138. doi: 10.1111/epi.17106. Epub 2021 Oct 22. PMID 34676542
- [Derived] Sullivan J, Perry MS, Wheless JW, Galer B, Gammaitoni A. Fenfluramine responder analyses and numbers needed to treat: Translating epilepsy trial data into clinical practice. Eur J Paediatr Neurol. 2021 Mar;31:10-14. doi: 10.1016/j.ejpn.2021.01.005. Epub 2021 Jan 22. PMID 33540241
- [Derived] Lagae L, Sullivan J, Knupp K, Laux L, Polster T, Nikanorova M, Devinsky O, Cross JH, Guerrini R, Talwar D, Miller I, Farfel G, Galer BS, Gammaitoni A, Mistry A, Morrison G, Lock M, Agarwal A, Lai WW, Ceulemans B; FAiRE DS Study Group. Fenfluramine hydrochloride for the treatment of seizures in Dravet syndrome: a randomised, double-blind, placebo-controlled trial. Lancet. 2019 Dec 21;394(10216):2243-2254. doi: 10.1016/S0140-6736(19)32500-0. Epub 2019 Dec 17. PMID 31862249

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study 1501 started to enroll participants in January 2016 and concluded in July 2020.
  The study 1502 started to enroll participants in July 2016 and concluded in July 2020. The consolidated results of Study 1 and Study 3 are included in this record. The Participant Flow refers to the Randomized Population.
Pre-assignment Details: Due to slow enrollment into both trials, the databases for the two trials were combined. The first 72 enrolled participants from ZX008-1501 and first 47 from ZX008-1502 were combined for an analysis and reported as Study 1, whereas the final 55 participants from ZX008- 1501 and the final 88 from ZX008-1502 were combined and reported as Study 3.
Groups:
- Study 1: Placebo: Participants received matching placebo as an oral solution, twice a day (bid) in equally divided doses with food for up to approximately 16 weeks. Study 1 is the merged analysis of 2 identical (ZX008-1501 and ZX008-1502) studies.
- Study 1: ZX008 0.2 mg/kg/Day: Participants received ZX008 0.2 milligram per kilogram per day (mg/kg/day) as an oral solution, bid, in equally divided doses with food for up to approximately 16 weeks. Study 1 is the merged analysis of 2 identical (ZX008-1501 and ZX008-1502) studies.
- Study 1: ZX008 0.8 mg/kg/Day: Participants received ZX008 0.8 mg/kg/day as an oral solution, bid, in equally divided doses with food for up to approximately 16 weeks. Study 1 is the merged analysis of 2 identical (ZX008-1501 and ZX008-1502) studies.
- Study 3: Placebo: Participants received matching placebo as an oral solution, bid, in equally divided doses with food for up to approximately 16 weeks. Study 3 is the merged analysis of 2 identical (ZX008-1501 and ZX008-1502) studies.
- Study 3: ZX008 0.2 mg/kg/Day: Participants received ZX008 0.2 mg/kg/day as an oral solution, bid, in equally divided doses with food for up to approximately 16 weeks. Study 3 is the merged analysis of 2 identical (ZX008-1501 and ZX008-1502) studies.
- Study 3: ZX008 0.8 mg/kg/Day: Participants received ZX008 0.8 mg/kg/day as an oral solution, bid, in equally divided doses with food for up to approximately 16 weeks. Study 3 is the merged analysis of 2 identical (ZX008-1501 and ZX008-1502) studies.
Period: Overall Study
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Started | 40 | 39 | 40 | 48 | 46 | 49
Completed | 37 | 39 | 34 | 43 | 45 | 46
Not Completed | 3 | 0 | 6 | 5 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 5 | 1 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refers to the Randomized population which included all participants randomized to receive study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day | Total
Number analyzed (Participants) | 40 | 39 | 40 | 48 | 46 | 49 | 262
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.2 (5.10) | 9.0 (4.52) | 8.8 (4.41) | 9.0 (4.29) | 9.6 (4.42) | 9.5 (5.29) | 9.2 (4.65)
Age, Customized [Count of Participants; unit: Participants]
  24 Months - <12 Years | 27 | 28 | 31 | 31 | 30 | 30 | 177
  12 - < 18 Years | 10 | 11 | 7 | 17 | 15 | 16 | 76
  18 - < 65 Years | 3 | 0 | 2 | 0 | 1 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 19 | 21 | 22 | 27 | 125
  Male | 21 | 22 | 21 | 27 | 24 | 22 | 137
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31 | 33 | 34 | 36 | 37 | 34 | 205
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Asian | 4 | 2 | 1 | 7 | 5 | 8 | 27
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Other | 2 | 1 | 1 | 4 | 2 | 3 | 13
  Not Reported | 2 | 2 | 4 | 1 | 0 | 1 | 10
  Unknown | 0 | 0 | 0 | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Mean Convulsive Seizures Frequency (MCSF) to the Combined Titration and Maintenance Periods (T+M) in Participants Receiving ZX008 0.8 mg/kg/Day Compared to Placebo
Description: Monthly (28 day) convulsive seizure frequency (CSF) was based on electronic diary data obtained for each participant. Convulsive seizures included hemiclonic, focal with clear observable motor signs, generalized tonic clonic, secondarily generalized tonic clonic, tonic, clonic, and drop seizures (tonic/atonic). The number of convulsive seizures reported during the entire time interval was divided by the number of nonmissing diary days and the result was then multiplied by 28 to get a 28-day CSF.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) plus Maintenance Period (12 weeks)]
Population: The modified intent-to-treat (mITT) population included all randomized participants who received at least 1 dose of ZX008 or placebo and for whom at least 1 week of diary data were available.
Measure: Mean (Standard Deviation); unit: seizure frequency per 28 days
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 40 | 48 | 48
seizure frequency per 28 days | -6.71 (24.263) | -13.11 (25.500) | 1.54 (21.966) | -3.54 (124.132)
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: ZX008 0.8 mg/kg/Day; Test type: Superiority; Percentage difference from Placebo = 62.29, 95% CI 2-sided [47.72 to 72.80] — Estimate was obtained from the LSMeans on the log scale as follows: 100 x [1 - exp(LS mean active - LS mean placebo)
Statistical Analysis 2: Comparison: Study 3: Placebo vs Study 3: ZX008 0.8 mg/kg/Day; Test type: Superiority; Percentage difference from Placebo = 64.75, 95% CI 2-sided [51.85 to 74.19] — Estimate was obtained from the LSMeans on the log scale as follows: 100 x [1 - exp(LS mean active - LS mean placebo)

2. Secondary Outcome: Change From Baseline in the Mean Convulsive Seizures Frequency to the Combined Titration and Maintenance Period (T+M) in Participants Receiving ZX008 0.2 mg/kg/Day Compared to Placebo
Description: as for outcome 1
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) plus Maintenance Period (12 weeks)]
Population: The mITT population included all randomized participants who received at least 1 dose of ZX008 or placebo and for whom at least 1 week of diary data were available.
Measure: Mean (Standard Deviation); unit: seizure frequency per 28 days
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 48 | 46
seizure frequency per 28 days | -6.71 (24.263) | -18.81 (90.640) | 1.54 (21.966) | -5.89 (84.735)
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: ZX008 0.2 mg/kg/Day; Test type: Superiority; Percentage difference from Placebo = 32.43, 95% CI 2-sided [6.19 to 51.33] — Estimate was obtained from the LSMeans on the log scale as follows: 100 x [1 - exp(LS mean active - LS mean placebo)
Statistical Analysis 2: Comparison: Study 3: Placebo vs Study 3: ZX008 0.2 mg/kg/Day; Test type: Superiority; Percentage difference from Placebo = 49.88, 95% CI 2-sided [31.31 to 63.43] — Estimate was obtained from the LSMeans on the log scale as follows: 100 x [1 - exp(LS mean active - LS mean placebo)

3. Secondary Outcome: Percentage of Participants Who Achieved Greater Than or Equal to 25% (≥25%) Reduction in Convulsive Seizure Frequency in Each ZX008 Treatment Arm Compared to Placebo From Baseline During the Titration and Maintenance Period
Description: Convulsive seizures included hemiclonic, focal with clear observable motor signs, generalized tonic clonic, secondarily generalized tonic clonic, tonic, clonic, and drop seizures (tonic/atonic). A responder was a participant who experienced a 25% or greater reduction in convulsive seizure frequency per 28 days during Titration and Maintenance Period.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) plus Maintenance Period (12 weeks)]
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 40 | 48 | 46 | 48
percentage of participants | 35.0 | 66.7 | 90.0 | 27.1 | 71.7 | 83.3

4. Secondary Outcome: Percentage of Participants Who Achieved a ≥50% Reduction in Convulsive Seizure Frequency in Each ZX008 Treatment Arm Compared to Placebo From Baseline During the Titration and Maintenance Period
Description: Convulsive seizures included hemiclonic, focal with clear observable motor signs, generalized tonic clonic, secondarily generalized tonic clonic, tonic, clonic, and drop seizures (tonic/atonic). A responder was a participant who experienced a 50% or greater reduction in convulsive seizure frequency per 28 days during Titration and Maintenance Period.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) plus Maintenance Period (12 weeks)]
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 40 | 48 | 46 | 48
percentage of participants | 12.5 | 38.5 | 67.5 | 6.3 | 45.7 | 72.9
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: ZX008 0.2 mg/kg/Day; Test type: Superiority; p = 0.009, Regression, Logistic; Odds Ratio (OR) = 4.773, 95% CI 2-sided [1.475 to 15.450]
Statistical Analysis 2: Comparison: Study 1: Placebo vs Study 1: ZX008 0.8 mg/kg/Day; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 14.960, 95% CI 2-sided [4.484 to 49.915]
Statistical Analysis 3: Comparison: Study 3: Placebo vs Study 3: ZX008 0.2 mg/kg/Day; Test type: Superiority; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 13.4, 95% CI 2-sided [3.6 to 49.8]
Statistical Analysis 4: Comparison: Study 3: Placebo vs Study 3: ZX008 0.8 mg/kg/Day; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 53.3, 95% CI 2-sided [12.9 to 220.5]

5. Secondary Outcome: Percentage of Participants Who Achieved a ≥75% Reduction in Convulsive Seizure Frequency in Each ZX008 Treatment Arm Compared to Placebo From Baseline During the Titration and Maintenance Period
Description: Convulsive seizures included hemiclonic, focal with clear observable motor signs, generalized tonic clonic, secondarily generalized tonic clonic, tonic, clonic, and drop seizures (tonic/atonic). A responder was a participant who experienced a 75% or greater reduction in convulsive seizure frequency per 28 days during Titration and Maintenance Period.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) plus Maintenance Period (12 weeks)]
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 40 | 48 | 46 | 48
percentage of participants | 2.5 | 23.1 | 50.0 | 4.2 | 28.3 | 47.9

6. Secondary Outcome: Percentage of Participants Who Achieved a 100% Reduction in Convulsive Seizure Frequency in Each ZX008 Treatment Arm Compared to Placebo From Baseline During the Titration and Maintenance Period
Description: Convulsive seizures included hemiclonic, focal with clear observable motor signs, generalized tonic clonic, secondarily generalized tonic clonic, tonic, clonic, and drop seizures (tonic/atonic). A responder was a participant who experienced a 100% reduction in convulsive seizure frequency per 28 days during Titration and Maintenance Period.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) plus Maintenance Period (12 weeks)]
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 40 | 48 | 46 | 48
percentage of participants | 0 | 7.7 | 7.5 | 0 | 0 | 12.5

7. Secondary Outcome: Longest Convulsive Seizure-free Interval in Each ZX008 Treatment Arm Compared to Placebo During the Titration and Maintenance Period
Description: The longest interval between convulsive seizures was calculated over the entire Titration and Maintenance Period and was derived as the maximum of the number of days between consecutive convulsive seizures.
Time Frame: During 14 weeks Titration (2 weeks) and Maintenance Period (12 weeks) (average of 99 days)
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 40 | 48 | 46 | 48
days | 9.50 [2.0 to 23.0] | 15.00 [3.0 to 106.0] | 25.00 [2.0 to 97.0] | 10 [2 to 65] | 18.5 [2 to 100] | 30 [2 to 104]
Statistical Analysis 1: Comparison: Study 1: Placebo vs Study 1: ZX008 0.2 mg/kg/Day; Test type: Superiority; p = 0.035, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Study 1: Placebo vs Study 1: ZX008 0.8 mg/kg/Day; Test type: Superiority; p < 0.001, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Study 3: Placebo vs Study 3: ZX008 0.2 mg/kg/Day; Test type: Superiority; p = 0.0002, Wilcoxon rank sum test; Comparing active with placebo
Statistical Analysis 4: Comparison: Study 3: Placebo vs Study 3: ZX008 0.8 mg/kg/Day; Test type: Superiority; p < 0.0001, Wilcoxon rank sum test

8. Secondary Outcome: Number of Convulsive Seizure-free Days in Each ZX008 Treatment Arm Compared to Placebo During the Titration and Maintenance Period
Description: A convulsive seizure free day was defined as a day for which diary data are available and no convulsive seizures were reported. Convulsive seizure free days were taken from the electronic diary data.
Time Frame: During 14 weeks Titration (2 weeks) and Maintenance Period (12 weeks) (average of 99 days)
Population: as for outcome 2
Measure: Median (Full Range); unit: seizure free days
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 40 | 48 | 46 | 48
seizure free days | 15.14 [1.1 to 25.6] | 20.86 [2.2 to 28.0] | 24.43 [1.0 to 28.0] | 20.20 [1.4 to 27.1] | 23.36 [0.8 to 27.7] | 25.33 [0.3 to 28.0]

9. Secondary Outcome: Change From Baseline in Non-convulsive Seizure Frequency to the Combined Titration and Maintenance Period in Each ZX008 Treatment Arm Compared to Placebo
Description: Non-convulsive seizures included focal without clear observable motor signs, absence or atypical absence, myoclonic and atonic. The number of non-convulsive seizures reported during the entire time interval was divided by the number of nonmissing diary days and the result was then multiplied by 28 to get a 28-day non-convulsive seizure frequency.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) plus Maintenance Period (12 weeks)]
Population: The mITT population included all randomized participants who received at least 1 dose of ZX008 or placebo and for whom at least 1 week of diary data were available. Here, number of participants analyzed included those participants who were evaluable for the assessment.
Measure: Median (Full Range); unit: seizure frequency per 28 days
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 21 | 23 | 24 | 26 | 25 | 30
seizure frequency per 28 days | -9.38 [-198.8 to 1886.1] | -4.85 [-1940.8 to 192.3] | -20.06 [-2064.8 to 9.4] | -0.68 [-160.0 to 1313.1] | -0.67 [-138.7 to 111.3] | -4.35 [-1410.6 to 107.5]

10. Secondary Outcome: Change From Baseline in Convulsive + Non-convulsive Seizure Frequency to the Combined Titration and Maintenance Period in Each ZX008 Treatment Arm Compared to Placebo
Description: Total seizure frequency were defined as the combination of convulsive and non-convulsive seizures. Convulsive seizures included hemiclonic, focal with clear observable motor signs, generalized tonic clonic, secondarily generalized tonic clonic, tonic, clonic, and drop seizures (tonic/atonic). Non-convulsive seizures included focal without clear observable motor signs, absence or atypical absence, myoclonic and atonic. The seizure frequency was based on electronic diary data obtained for each participant. The number of all seizures reported during the entire time interval was divided by the number of nonmissing diary days and the result was then multiplied by 28 to get a 28-day convulsive or non-convulsive seizure frequency.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) plus Maintenance Period (12 weeks)]
Population: as for outcome 2
Measure: Median (Full Range); unit: seizure frequency per 28 days
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 40 | 48 | 46 | 48
seizure frequency per 28 days | -4.45 [-198.4 to 1850.1] | -7.40 [-1955.1 to 187.1] | -22.95 [-2069.3 to 44.5] | -1.09 [-160.1 to 1310.5] | -6.54 [-153.0 to 525.9] | -11.39 [-1504.8 to 791.4]

11. Secondary Outcome: Percentage of Participants With Rescue Medication Usage in Each ZX008 Treatment Arm Compared to Placebo During the Titration and Maintenance Period
Description: Rescue medication was administered according to each participant's usual or prescribed regimen consisting of 1 or more medications. The usage of rescue medication (number of days and number of medications used per seizure episode) was based on electronic diary data obtained for each participant. The number of days rescue medication was taken (normalized to 28 days) was calculated for each participant. Multiple medications taken on the same day were counted once for that day.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) plus Maintenance Period (12 weeks)]
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 40 | 48 | 46 | 48
percentage of participants | 77.5 | 59.0 | 45.0 | 60.4 | 65.2 | 47.9

12. Secondary Outcome: Percentage of Participants With Hospitalization and Healthcare Resource Utilization to Treat Seizures in Each ZX008 Treatment Arm Compared to Placebo During Study
Description: Participants who utilized medical center care to treat a seizure during the study were reported.
Time Frame: During 14 weeks Titration (2 weeks) and Maintenance Period (12 weeks) (average of 99 days)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 40 | 48 | 46 | 48
percentage of participants | 22.5 | 17.9 | 15.0 | 12.5 | 19.6 | 14.6

13. Secondary Outcome: Percentage of Participants With Status Epilepticus (SE) in Each ZX008 Treatment Arm Compared to Placebo During the Titration and Maintenance Period
Description: The participants who either had SE episode recorded as an adverse event (AE) during treatment or a seizure greater than 10 minutes were reported for each treatment group. Additionally, a single participant who may had more than one episode of SE, and an episode of SE recorded as both an AE and as a seizure longer than 10 minutes was counted as a single event.
Time Frame: During 14 weeks Titration (2 weeks) and Maintenance Period (12 weeks) (average of 99 days)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 40 | 48 | 46 | 48
percentage of participants | 27.5 | 28.2 | 35.0 | 16.7 | 19.6 | 25.0

14. Secondary Outcome: Distribution of Duration of Convulsive Seizures (in Percentage) in Each ZX008 Treatment Arm Compared to Placebo at Baseline and During the Titration and Maintenance Period
Description: Duration of single convulsive seizures during the Baseline and the duration over the Titration and Maintenance Period were reported by treatment group using categories as <2 minutes, 2 to 10 minutes and > 10 minutes as collected in the seizure diary.
Time Frame: At Baseline and 14 weeks of Titration (2 weeks) and Maintenance Period (12 weeks)
Population: as for outcome 2
Measure: Number; unit: percentage of seizures
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 40 | 48 | 46 | 48
percentage of seizures
  <2 min (Baseline) | 69.28 | 64.13 | 71.61 | 64.21 | 63.90 | 74.11
  2-10 min (Baseline) | 26.86 | 34.95 | 24.22 | 34.83 | 33.66 | 22.78
  >10 min (Baseline) | 3.86 | 0.93 | 4.17 | 0.96 | 2.45 | 3.10
  <2 min (Titration + Maintenance Period) | 71.31 | 71.59 | 72.27 | 65.84 | 63.45 | 84.67
  2-10 min (Titration + Maintenance Period) | 26.31 | 25.61 | 22.91 | 33.74 | 31.34 | 13.71
  >10 min (Titration + Maintenance Period) | 2.38 | 2.79 | 4.82 | 0.43 | 5.22 | 1.62

15. Secondary Outcome: Percentage of Participants With Clinical Global Impression - Improvement (CGI-I) Rating Score, as Assessed by the Principal Investigator in Each ZX008 Treatment Arm Compared to Placebo
Description: CGI-I scale measures improvement in the participant's clinical status from Baseline. The severity of a participant's condition was rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse), as follows: 1-very much improved,2-much improved, 3-minimally improved, 4- no change, 5-minimally worse, 6-much worse and 7-very much worse. The Principal Investigator rated their global impression of the participant's condition during the study.
Time Frame: At Visit 6 (Day 15), 8 (Day 43), 10 (Day 71) and 12 (Day 99)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 40 | 48 | 46 | 48
percentage of participants
  1 = Very much improved (Visit 6) | 5.0 | 23.1 | 17.5 | 4.2 | 21.7 | 16.7
  2 = Much improved (Visit 6) | 12.5 | 12.8 | 25.0 | 2.1 | 21.7 | 27.1
  3 = Minimally improved (Visit 6) | 20.0 | 20.5 | 20.0 | 27.1 | 17.4 | 27.1
  4 = No change (Visit 6) | 40.0 | 25.6 | 17.5 | 54.2 | 26.1 | 12.5
  5 = Minimally worse (Visit 6) | 5.0 | 7.7 | 5.0 | 4.2 | 2.2 | 2.1
  6 = Much worse (Visit 6) | 0 | 0 | 2.5 | 0 | 0 | 4.2
  7 = Very much worse (Visit 6) | 0 | 0 | 0 | 0 | 0 | 0
  1 = Very much improved (Visit 8) | 0 | 5.1 | 17.5 | 4.2 | 17.4 | 29.2
  2 = Much improved (Visit 8) | 12.5 | 30.8 | 37.5 | 6.3 | 10.9 | 31.3
  3 = Minimally improved (Visit 8) | 30.0 | 20.5 | 10.0 | 16.7 | 26.1 | 14.6
  4 = No change (Visit 8) | 30.0 | 17.9 | 10.0 | 50.0 | 34.8 | 8.3
  5 = Minimally worse (Visit 8) | 5.0 | 5.1 | 0 | 4.2 | 0 | 4.2
  6 = Much worse (Visit 8) | 2.5 | 5.1 | 2.5 | 2.1 | 0 | 0
  7 = Very much worse (Visit 8) | 0 | 0 | 2.5 | 0 | 0 | 0
  1 = Very much improved (Visit 10) | 2.5 | 17.9 | 20.0 | 4.2 | 15.2 | 35.4
  2 = Much improved (Visit 10) | 7.5 | 17.9 | 47.5 | 10.4 | 19.6 | 18.8
  3 = Minimally improved (Visit 10) | 30.0 | 25.6 | 5.0 | 12.5 | 26.1 | 16.7
  4 = No change (Visit 10) | 35.0 | 28.2 | 7.5 | 60.4 | 28.3 | 4.2
  5 = Minimally worse (Visit 10) | 10.0 | 7.7 | 0 | 0 | 0 | 0
  6 = Much worse (Visit 10) | 0 | 2.6 | 0 | 0 | 0 | 2.1
  7 = Very much worse (Visit 10) | 0 | 0 | 0 | 0 | 0 | 0
  1 = Very much improved (Visit 12) | 2.5 | 12.8 | 27.5 | 4.2 | 8.7 | 33.3
  2 = Much improved (Visit 12) | 7.5 | 28.2 | 35.0 | 4.2 | 28.3 | 31.3
  3 = Minimally improved (Visit 12) | 30.0 | 17.9 | 15.0 | 16.7 | 21.7 | 10.4
  4 = No change (Visit 12) | 47.5 | 28.2 | 12.5 | 58.3 | 28.3 | 16.7
  5 = Minimally worse (Visit 12) | 2.5 | 10.3 | 0 | 6.3 | 10.9 | 6.3
  6 = Much worse (Visit 12) | 2.5 | 2.6 | 0 | 0 | 0 | 0
  7 = Very much worse (Visit 12) | 0 | 0 | 2.5 | 0 | 0 | 0

16. Secondary Outcome: Percentage of Participants With Clinical Global Impression - Improvement Rating Score, as Assessed by the Parent/Caregiver in Each ZX008 Treatment Arm Compared to Placebo
Description: CGI-I scale measures improvement in the participant's clinical status from Baseline. The severity of a participant's condition was rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse), as follows: 1-very much improved,2-much improved, 3-minimally improved, 4- no change, 5-minimally worse, 6-much worse and 7-very much worse. The Parent/Caregiver rated their global impression of the participant's condition during the study.
Time Frame: At Visit 6 (Day 15), 8 (Day 43), 10 (Day 71) and 12 (Day 99)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 40 | 48 | 46 | 48
percentage of participants
  1 = Very much improved (Visit 6) | 2.5 | 17.9 | 15.0 | 6.3 | 13.0 | 16.7
  2 = Much improved (Visit 6) | 22.5 | 20.5 | 27.5 | 2.1 | 23.9 | 31.3
  3 = Minimally improved (Visit 6) | 12.5 | 28.2 | 22.5 | 25.0 | 26.1 | 31.3
  4 = No change (Visit 6) | 45.0 | 12.8 | 20.0 | 45.8 | 19.6 | 2.1
  5 = Minimally worse (Visit 6) | 2.5 | 7.7 | 2.5 | 10.4 | 2.2 | 6.3
  6 = Much worse (Visit 6) | 5.0 | 2.6 | 7.5 | 2.1 | 2.2 | 2.1
  7 = Very much worse (Visit 6) | 0 | 0 | 2.5 | 0 | 0 | 2.1
  1 = Very much improved (Visit 8) | 0 | 15.4 | 20.0 | 4.2 | 6.5 | 39.6
  2 = Much improved (Visit 8) | 15.0 | 25.6 | 37.5 | 8.3 | 30.4 | 29.2
  3 = Minimally improved (Visit 8) | 25.0 | 25.6 | 15.0 | 20.8 | 28.3 | 14.6
  4 = No change (Visit 8) | 20.0 | 12.8 | 5.0 | 47.9 | 17.4 | 6.3
  5 = Minimally worse (Visit 8) | 15.0 | 10.3 | 2.5 | 6.3 | 6.5 | 0
  6 = Much worse (Visit 8) | 2.5 | 5.1 | 5.0 | 4.2 | 2.2 | 2.1
  7 = Very much worse (Visit 8) | 0 | 0 | 2.5 | 4.2 | 0 | 0
  1 = Very much improved (Visit 10) | 2.5 | 20.5 | 35.0 | 2.1 | 8.7 | 41.7
  2 = Much improved (Visit 10) | 12.5 | 17.9 | 30.0 | 6.3 | 28.3 | 22.9
  3 = Minimally improved (Visit 10) | 22.5 | 20.5 | 7.5 | 25.0 | 26.1 | 8.3
  4 = No change (Visit 10) | 32.5 | 25.6 | 10.0 | 45.8 | 26.1 | 6.3
  5 = Minimally worse (Visit 10) | 12.5 | 7.7 | 0 | 6.3 | 0 | 4.2
  6 = Much worse (Visit 10) | 2.5 | 7.7 | 0 | 0 | 4.3 | 0
  7 = Very much worse (Visit 10) | 2.5 | 0 | 2.5 | 0 | 0 | 0
  1 = Very much improved (Visit 12) | 2.5 | 20.5 | 27.5 | 2.1 | 6.5 | 33.3
  2 = Much improved (Visit 12) | 7.5 | 20.5 | 27.5 | 6.3 | 28.3 | 29.2
  3 = Minimally improved (Visit 12) | 20.0 | 15.4 | 10.0 | 18.8 | 30.4 | 20.8
  4 = No change (Visit 12) | 35.0 | 20.5 | 15.0 | 50.0 | 13.0 | 4.2
  5 = Minimally worse (Visit 12) | 17.5 | 15.4 | 5.0 | 10.4 | 8.7 | 4.2
  6 = Much worse (Visit 12) | 7.5 | 7.7 | 5.0 | 2.1 | 4.3 | 2.1
  7 = Very much worse (Visit 12) | 0 | 0 | 2.5 | 0 | 2.2 | 2.1

17. Secondary Outcome: Change From Baseline to Day 99 in the Quality of Life in Childhood Epilepsy (QOLCE) Score to Measure Quality of Life in Each ZX008 Treatment Arm Compared to Placebo
Description: QOLCE is a low-burden parent/caregiver completed assessment that evaluates how epilepsy affects day-to day functioning of the participant in various life areas, including physical activities, well being, cognition, social activities, behavior, and general health. QOLCE scores items on 16 subscales with possible 5-point response for each, where scores of 5 was best possible response and 1 was worst possible response. Item scores were then transformed to a 0-100 scale as follows: 1-0, 2-25, 3-50, 4-75, 5-100. A score for each participant for each subscale was calculated by averaging that participant's responses to each item in the subscale. Subscale scores per participant were averaged to obtain an overall QoL score for each participant. Higher the subscale and overall QoL scores, better the response.
Time Frame: From Baseline to Day 99
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 40 | 48 | 46 | 48
score on a scale | 1.5 (8.73) | 0.8 (11.77) | 5.8 (11.70) | 1.2 (9.01) | 6.1 (12.47) | 5.5 (13.22)

18. Secondary Outcome: Change From Baseline to Day 99 in the Overall Quality of Life Score From the Pediatric Quality of Life Inventory™ (PedsQL) Score in Each ZX008 Treatment Arm Compared to Placebo
Description: The Pediatric Quality of Life Inventory (PedsQL) is a pediatric modular measure of health related quality of life (QoL) completed by the parent/caregiver on behalf of the participant. It consisted of 23 items across 4 core scales that measure physical (8 items), emotional, social, and school functioning (5 items each). Each of the responses to the 23 items is initially scored on a 5-point Likert scale from 0 (Never) to 4 (Almost always). Scores are linearly transformed to a scale of 0 to 100, where 0=100, 1=75, 2=50, 3=25 and 4=0, and higher scores correspond to better health-related QoL. The Overall Quality of Life is the average of all the items over the number of items answered on all the Scales.
Time Frame: From Baseline to Day 99
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 40 | 48 | 46 | 48
score on a scale | -1.6 (10.43) | 6.8 (11.25) | 5.9 (15.11) | 1.9 (13.26) | 4.2 (17.65) | 2.1 (14.73)

19. Secondary Outcome: Change From Baseline to Day 99 in the Total Score From PedsQL Family Impact Module Score in Each ZX008 Treatment Arm Compared to Placebo
Description: The PedsQL Family Impact measured the impact of pediatric chronic health conditions on parents and the family by measuring parent self-reported physical, emotional, social, and cognitive functioning, communication, worry, and family daily activities and relationships. There are a total of 36 items in the PedsQL: 6 items for Physical Functioning, 5 items each for Emotional Functioning, Cognitive Functioning and Worry, 4 for Social Functioning, 3 for Communication, 3 questions for Daily Activities, and 5 for Family Relationships. Each of the responses are initially scored on a 5-point Likert scale from 0 (Never) to 4 (Almost always) and then linearly transformed to a scale of 0 to 100, where 0=100, 1=75, 2=50, 3=25 and 4=0, and higher scores mean better health-related QoL.
Time Frame: From Baseline to Day 99
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 40 | 39 | 40 | 47 | 44 | 48
score on a scale | -4.4 (13.00) | 3.9 (9.44) | 5.4 (15.60) | 1.3 (14.88) | 0.7 (15.78) | 6.3 (14.64)

20. Secondary Outcome: Quality of Life (QoL) of the Parent/Caregiver Using the EQ- 5D-5L Scale in Each ZX008 Treatment Arm Compared to Placebo at Baseline and Day 99
Description: The EuroQOL-5 Dimensions-5 Levels scale produced by European QOL Group (EQ-5D-5L) health questionnaire is a health-related QOL instrument with 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The 5 dimensions of EQ-5D-5L health questionnaire were assessed on a Likert scale with 5 possible levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The categories "slight problems", "moderate problems", "severe problems" and "extreme problems" are collapsed into one response category "problems. The QOL of the parent/caregiver was assessed and percentage of participants was reported for each item.
Time Frame: At Baseline and Day 99
Population: The mITT population included all randomized participants who received at least 1 dose of ZX008 or placebo and for whom at least 1 week of diary data were available. Here, Number of participants analyzed included those participants who were evaluable for the assessment and 'n' (Number analyzed) signifies participants who were evaluable at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 39 | 37 | 39 | 42 | 43 | 45
percentage of participants
  Mobility- No problems (Baseline): number analyzed (Participants) | 39 | 34 | 39 | 40 | 33 | 35
  Mobility- No problems (Baseline) | 33.33 | 52.94 | 46.15 | 40.00 | 54.55 | 28.57
  Mobility- Problems (Baseline): number analyzed (Participants) | 39 | 34 | 39 | 40 | 33 | 35
  Mobility- Problems (Baseline) | 66.67 | 47.06 | 53.85 | 60.00 | 45.45 | 71.43
  Mobility- No problems (Day 99): number analyzed (Participants) | 35 | 37 | 37 | 42 | 43 | 45
  Mobility- No problems (Day 99) | 40.00 | 45.95 | 51.35 | 52.38 | 51.16 | 46.67
  Mobility- Problems (Day 99): number analyzed (Participants) | 35 | 37 | 37 | 42 | 43 | 45
  Mobility- Problems (Day 99) | 60.00 | 54.05 | 48.65 | 47.62 | 48.84 | 53.33
  Self-care - No problems (Baseline): number analyzed (Participants) | 39 | 34 | 39 | 40 | 33 | 35
  Self-care - No problems (Baseline) | 25.64 | 41.18 | 38.46 | 22.50 | 36.36 | 22.86
  Self-care - Problems (Baseline): number analyzed (Participants) | 39 | 34 | 39 | 40 | 33 | 35
  Self-care - Problems (Baseline) | 74.36 | 58.82 | 61.54 | 77.50 | 63.64 | 77.14
  Self-care - No problems (Day 99): number analyzed (Participants) | 35 | 37 | 37 | 42 | 43 | 45
  Self-care - No problems (Day 99) | 28.57 | 43.24 | 48.65 | 30.95 | 34.88 | 35.56
  Self-care - Problems (Day 99): number analyzed (Participants) | 35 | 37 | 37 | 42 | 43 | 45
  Self-care - Problems (Day 99) | 71.43 | 56.76 | 51.35 | 69.05 | 65.12 | 64.44
  Usual activities- No problems (Baseline): number analyzed (Participants) | 39 | 34 | 39 | 40 | 33 | 35
  Usual activities- No problems (Baseline) | 23.08 | 41.18 | 35.90 | 25.00 | 39.39 | 20.00
  Usual activities- Problems (Baseline): number analyzed (Participants) | 39 | 34 | 39 | 40 | 33 | 35
  Usual activities- Problems (Baseline) | 76.92 | 58.82 | 64.10 | 75.00 | 60.61 | 80.00
  Usual activities- No problems (Day 99): number analyzed (Participants) | 35 | 37 | 37 | 42 | 43 | 45
  Usual activities- No problems (Day 99) | 25.71 | 32.43 | 48.65 | 30.95 | 25.58 | 35.56
  Usual activities- Problems (Day 99): number analyzed (Participants) | 35 | 37 | 37 | 42 | 43 | 45
  Usual activities- Problems (Day 99) | 74.29 | 67.57 | 51.35 | 69.05 | 74.42 | 64.44
  Pain/discomfort- No problems (Baseline): number analyzed (Participants) | 39 | 34 | 39 | 40 | 33 | 35
  Pain/discomfort- No problems (Baseline) | 48.72 | 41.18 | 46.15 | 45.00 | 51.52 | 51.43
  Pain/discomfort- Problems (Baseline): number analyzed (Participants) | 39 | 34 | 39 | 40 | 33 | 35
  Pain/discomfort- Problems (Baseline) | 51.28 | 58.82 | 53.85 | 55.00 | 48.48 | 48.57
  Pain/discomfort- No problems (Day 99): number analyzed (Participants) | 35 | 37 | 37 | 42 | 43 | 45
  Pain/discomfort- No problems (Day 99) | 48.57 | 51.35 | 64.86 | 76.19 | 46.51 | 64.44
  Pain/discomfort- Problems (Day 99): number analyzed (Participants) | 35 | 37 | 37 | 42 | 43 | 45
  Pain/discomfort- Problems (Day 99) | 51.43 | 48.65 | 35.14 | 45.24 | 53.49 | 35.56
  Anxiety/depression- No problems (Baseline): number analyzed (Participants) | 39 | 34 | 39 | 40 | 33 | 35
  Anxiety/depression- No problems (Baseline) | 74.36 | 61.76 | 56.41 | 60.00 | 63.64 | 74.29
  Anxiety/depression- Problems (Baseline): number analyzed (Participants) | 39 | 34 | 39 | 40 | 33 | 35
  Anxiety/depression- Problems (Baseline) | 25.64 | 38.24 | 43.59 | 40.00 | 36.36 | 25.71
  Anxiety/depression- No problems (Day 99): number analyzed (Participants) | 35 | 37 | 37 | 42 | 43 | 45
  Anxiety/depression- No problems (Day 99) | 65.71 | 67.57 | 67.57 | 69.05 | 67.44 | 73.33
  Anxiety/depression- Problems (Day 99): number analyzed (Participants) | 35 | 37 | 37 | 42 | 43 | 45
  Anxiety/depression- Problems (Day 99) | 34.29 | 32.43 | 32.43 | 30.95 | 32.56 | 26.67

21. Secondary Outcome: Change From Baseline to Day 99 in Affective Symptoms of the Parent/Caregiver Using the Hospital Anxiety and Depression Scale (HADS) in Each ZX008 Treatment Arm Compared to Placebo
Description: The HADS is a tool that was validated to assess presence of anxiety or depression in an outpatient non-psychiatric population. The HADS a 14-item scale that generates ordinal data for 2 dimensions: 1) Anxiety (7 items), and 2) Depression (7 items). Each item has 4 possible answers rated 0 to 3, of which 0 = No distress and 3 = worst distress. All answers to the items for a dimension with their respective rating are added resulting in a range for each dimension from 0-21, out of which of 0-7 = normal; 8-10=borderline abnormal; 11-21=abnormal. Scores for the entire scale (emotional distress) range from 0 to 42, with higher scores indicating more distress.
Time Frame: From Baseline to Day 99
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 31 | 32 | 35 | 30 | 31 | 27
score on a scale
  Anxiety | -0.4 (2.68) | -0.8 (2.84) | -0.8 (3.33) | -0.6 (3.62) | 0.2 (3.89) | -0.7 (4.00)
  Depression | 0.8 (4.50) | 0.2 (4.52) | 0.1 (4.35) | -0.7 (3.80) | 2.0 (4.77) | -0.8 (4.03)
  Total emotional distress | 0.4 (6.45) | -0.6 (6.60) | -0.7 (6.82) | -1.2 (6.42) | 2.2 (7.52) | -1.5 (6.61)

22. Secondary Outcome: Maximum Observed Concentration of ZX008 Determined Directly From the Concentration Time Profile [Cmax] at Steady State
Description: Cmax is the maximum observed concentration determined directly from the concentration-time profile.
Time Frame: At Visit 8 (Day 43): pre-dose, 1, 2, and 4-6 hours postdose
Population: PK population for each study represents participants randomized to ZX008 and provided concentrations for use in the population PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 39 | 36 | 45 | 44
nanograms per milliliter (ng/mL) | 17.7 (32.5) | 67.9 (37.4) | 17.4 (32.3) | 64.5 (36.6)

23. Secondary Outcome: Area Under the Concentration Time Curve of ZX008 From Time Zero to Time 24 Hours [AUC0-24hours] at Steady State
Description: AUC0-24 is the area under the concentration time curve from time zero to 24 hours.
Time Frame: At Visit 8 (Day 43): pre-dose, 1, 2, and 4-6 hours postdose
Population: PK population for each study represents participants randomized to ZX008 and provided concentrations for use in the population PK analysis. PK samples at Visit 8 (Day 43) taken pre-dose to 6 hours post-dose were used to develop a population PK model. The model was utilized to generate plasma concentration-time curve over 24 hours at steady-state in study participants. AUC0-24 was calculated by numerical integration of the individual predicted concentration-time curve.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 39 | 36 | 45 | 44
nanogram*hour per milliliter (ng*h/mL) | 356 (37.0) | 1390 (41.3) | 348 (37.1) | 1290 (42.6)

24. Secondary Outcome: Time to Maximum Concentration [Tmax] of ZX008 at Steady State
Description: Tmax is the time to maximum concentration at steady state.
Time Frame: At Visit 8 (Day 43): pre-dose, 1, 2, and 4-6 hours postdose
Population: as for outcome 22
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 39 | 36 | 45 | 44
hours (h) | 2.90 [2.80 to 3.10] | 3.00 [2.70 to 3.20] | 2.90 [2.80 to 3.10] | 2.90 [2.70 to 3.20]

25. Secondary Outcome: Elimination Half-life [t1/2 Beta] of ZX008 at Steady State
Description: t1/2 beta is the elimination half-life.
Time Frame: At Visit 8 (Day 43): pre-dose, 1, 2, and 4-6 hours postdose
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (h)
Arm/Group | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 39 | 36 | 45 | 44
hours (h) | 18.4 (32.3) | 21.1 (51.8) | 18.1 (32.1) | 18.6 (42.2)

ADVERSE EVENTS:
Time Frame: From Titration Period until the Safety Follow-up Visit (up to Day 113)
Description: A Treatment emergent adverse event (TEAE) was defined as any AE that based on start date information occurred after the first dose of study drug. The safety population included all randomized participants who received at least 1 dose of ZX008 or placebo.
Arm/Group | Study 1: Placebo | Study 1: ZX008 0.2 mg/kg/Day | Study 1: ZX008 0.8 mg/kg/Day | Study 3: Placebo | Study 3: ZX008 0.2 mg/kg/Day | Study 3: ZX008 0.8 mg/kg/Day
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39 | 0/40 | 1/48 | 0/46 | 0/48
Serious Adverse Events (participants affected / at risk) | 4/40 | 4/39 | 5/40 | 2/48 | 3/46 | 3/48
Other Adverse Events (participants affected / at risk) | 22/40 | 35/39 | 36/40 | 37/48 | 41/46 | 41/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study 1: Placebo (N=40) | Study 1: ZX008 0.2 mg/kg/Day (N=39) | Study 1: ZX008 0.8 mg/kg/Day (N=40) | Study 3: Placebo (N=48) | Study 3: ZX008 0.2 mg/kg/Day (N=46) | Study 3: ZX008 0.8 mg/kg/Day (N=48)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden unexplained death in epilepsy (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study 1: Placebo (N=40) | Study 1: ZX008 0.2 mg/kg/Day (N=39) | Study 1: ZX008 0.8 mg/kg/Day (N=40) | Study 3: Placebo (N=48) | Study 3: ZX008 0.2 mg/kg/Day (N=46) | Study 3: ZX008 0.8 mg/kg/Day (N=48)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 12 (14) | 7 (7) | 4 (4) | 7 (8) | 7 (7)
Vomiting (Gastrointestinal disorders) | 4 (5) | 4 (5) | 3 (3) | 3 (4) | 0 (0) | 3 (3)
Fatigue (General disorders) | 1 (1) | 4 (4) | 4 (4) | 1 (1) | 3 (3) | 5 (5)
Pyrexia (General disorders) | 8 (12) | 7 (12) | 2 (3) | 4 (5) | 5 (7) | 9 (11)
Nasopharyngitis (Infections and infestations) | 5 (6) | 4 (4) | 7 (8) | 5 (8) | 4 (7) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (7) | 8 (13) | 0 (0) | 2 (3) | 3 (4) | 4 (5)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 11 (13) | 8 (8)
Blood pressure diastolic increased (Investigations) | 1 (2) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 1 (1)
Echocardiogram abnormal (Investigations) | 5 (5) | 7 (7) | 9 (13) | 5 (5) | 11 (11) | 8 (8)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 8 (11) | 14 (15) | 3 (3) | 12 (12) | 18 (22)
Lethargy (Nervous system disorders) | 2 (2) | 4 (6) | 7 (8) | 2 (2) | 1 (1) | 3 (4)
Somnolence (Nervous system disorders) | 3 (4) | 6 (6) | 3 (3) | 5 (5) | 5 (6) | 10 (10)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Croup infectious (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 1 (3)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 3 (4) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Blood pressure systolic increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood prolactin increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 3 (3) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Weight decreased (Investigations) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Ataxia (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Drooling (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 3 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 4 (4) | 3 (5) | 2 (4) | 1 (1) | 0 (0) | 1 (1)
Seizure cluster (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 6 (6)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 2 (2)
Enuresis (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Negativism (Psychiatric disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 4 (4)

LIMITATIONS AND CAVEATS:
The full results posting consists of the pooled analysis 1 and 2 of the studies with study ID ZX008-1501 and ZX008-1502. Pooled analysis 1 is referenced as Study 1 in the respective statistical analysis plan (SAP) and corresponding clinical study report (CSR). Pooled analysis 2 is referenced as Study 2 in the respective SAP and, due to the timing of regulatory submissions, Study 3 in the corresponding CSR and in this results posting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/27/NCT02682927/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT02682927/SAP_001.pdf